CLINICAL TRIAL: NCT03230032
Title: RCT of Feeding Intervention With Pacifier Activated Device and Mother's Voice in Infants at High-risk for Cerebral Palsy.
Brief Title: Pacifier Activated Device and Mother's Voice in Infants at High-risk for Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: Cerebral Palsy Alliance (Other)
Responsible Party: Principal Investigator, Kristen Benninger, MD, Principle Investigator, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB16-00862
Record Dates: First submitted 2017-06-22; First posted 2017-07-26 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Infant Development; Infant,Premature; Hydrocephalus; Neonatal Encephalopathy; Infarction; PVL; Thrombosis; Intraventricular Hemorrhage
MeSH Terms: conditions — Premature Birth; Hydrocephalus; Infarction; Thrombosis

STUDY DESIGN:
Intervention Model Description: There participants will be randomized to two groups: PAL (pacifier and mother's voice provided contingently on sucking behavior) or Sounds of Love (listening to mother's voice not contingent upon sucking behavior on the pacifier, but pacifier available, per standard of care). To allow for high repetitiveness of the treatment, participants in both groups will receive 2 daily 15-min sessions of the intervention or control treatments for a total of 20 sessions. Sessions occur 15-30 min prior to feeding.
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intervention Group (Experimental): Sessions will use a pacifier-activated device (PAL) system. The device sensor attaches to a routinely-used pacifier and measures timing and pressure of the sucks. If the infant reaches the preset suck pressure, he receives 10 seconds of mother's voice. The receiver/speaker box controls the volume to < 65dB on scale C. PAM will be set to the lowest settings for the first session. Using sensor measurements, the therapist will increase the threshold for number of sucks and strength once the infant produces three consecutive sucks above current level and continue per protocol.
  Interventions: Device: pacifier-activated device
- Control Group (No Intervention): Infants will receive 2 daily 15-min listening sessions of mother's voice recording, contiguous but not simultaneous with PAM NNS sessions without suck-contingent reinforcement (no voice).

INTERVENTIONS:
Device: pacifier-activated device — The utilization of the pacifier-activated-music player combines the sound of the mother's voice with a pacifier routinely used with each patient during their inpatient NICU stay
  Other Names: PAL
  Arms: Intervention Group

SUMMARY:
The study seeks to determine the efficacy of non-nutritive suck (NNS) training using a pacifier-activated device (PAM) with mothers' voice to condition suck-strength and rhythmicity, in improving the feeding and developmental outcomes of infants at high-risk for CP.

DETAILED DESCRIPTION:
Poor neuromotor and sensory function of the aerodigestive system in children with CP often originates in the neonatal period, when they are still classified as "high-risk for CP". Characteristic neuroimaging abnormalities including severe intraventricular (IVH) hydrocephalus and periventricular leukomalacia (PVL), stroke or ischemia with lesions affect the posterior limb of the internal capsule are strong Indicators of high-risk for CP, especially when combined with abnormal General Movements Assessment (Guidelines for Early Detection of CP; Stockholm, 2016). Early intervention, when plasticity is greatest has the largest impact on functional recovery in CP. While intervening in infancy involves treating some infants who will not develop CP, the goal is to establish new neuronal connections and functional patterns before less efficient adaptations can occur. However, no current interventions target the oral-motor dysfunction of infants at high-risk for CP, before their discharge from the NICU.

Evidence for behavioral interventions in feeding disorders for children with CP ranges from insufficient to moderate, with a clear need for rigorous studies. In healthy preterm and late-preterm infants, oromotor practice opportunities such as non-nutritive suck (NNS) are safe and promote effective suck-swallow-breathe patterns, with decreased time to achieving oral feeds. While NNS opportunities are frequent in most NICUs, they must be adapted for effectiveness in infants at high-risk for CP. Motor learning in these infants must incorporate repetitive, self-initiated and task-directed activities. Learning is optimized when contingent on feedback, such as positive reinforcement.

NNS training (rather than simple exposure) has been implemented successfully using rhythmic sound of mother's voice singing contingent upon suck strength and pattern, as detected by a pacifier-sensor device (Pacifier-activated music; PAM) in an cohort of predominantly healthy preterm infants. An RCT demonstrated that NNS-trained infants had feeding tubes removed one week earlier than controls, with fewer aspiration events and feeding difficulties in infancy. The intervention was promising in the dozen infants with significant neural injury. Following this preliminary data, this study seeks to further determining the efficacy of non-nutritive suck (NNS) training using a pacifier-activated device (PAM) with mothers' voice to condition suck-strength and rhythmicity, in improving the feeding and developmental outcomes of infants at high-risk for CP.

ELIGIBILITY:
Inclusion Criteria:

* PMA at enrollment >32 6/7 and <42 AND
* Diagnoses of Grade III/IV IVH, hydrocephalus or PVL, neonatal encephalopathy or thrombosis/infarct with involvement of the posterior limb of the internal capsule OR
* Abnormal GMA by certified study staff and masked gold-standard reading

Exclusion Criteria: Infants cannot be

* on assisted ventilation
* receiving more than 50% of their feeds orally averaged over the 72 hours prior to study start
* receiving less than 50% of their feeds enterally
* receiving enteral feed for greater than 60 min.
* considered medically unsafe to feed orally by the medical or feeding team as defined by unit/clinical protocol

Ages: 32 Weeks to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 130 (Actual)
Dates: Start 2017-06-09 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Oral Feeding Efficiency | Twelve months
  Continuous measure of suck strength and suck rate during non-nutritive suck via PAM sensor, as well as suck burst pattern and average oral feeding volumes.

SECONDARY OUTCOMES:
HINE | 3-4 month and 12 month assessments
  Hammersmith Infant Neurologic Exam (HINE): standardized and scored neurological examination for infants 2-24 months; sequential use allows identification of early signs of CP and other neuromotor disorders. It includes 26 items assessing cranial nerve function, posture, quality and quantity of movements, muscle tone, and reflexes and reactions. Each item is scored individually (0, 1, 2 or 3), with a sum score of all individual items (range: 0-78). The maximum score for any one item is a score of 3 and the minimum is a score of 0.
Bayley-III | 3-4 months and 12 month assessments
  Bayley Scales of Infant and Toddler Development (Bailey-III): Standardized comprehensive assessment tool for assessing child development in children one month to 42 months old. Subtests assess adaptive behavior, cognitive, language, motor, and social-emotional domains. The highest possible scaled score on each subtest is 19, and the lowest possible score is 1. Scores from 8 to 12 are considered average. Composite scores are derived for each domain from sums of subtest scaled scores. Composite scores range from 40-160.
Oral feeding development questionnaire | 3-4 months and 12 month assessments
  Age-calibrated questionnaire (< or > 6 months) in the American Speech-Language-Hearing Association evidence maps for evaluation of feeding problems.
NOMAS | 33-41 weeks PMA and 35-43 weeks PMA
  Neonatal Oral-Motor Assessment Scale (NOMAS): A tool for the evaluation of neonatal nutritive sucking patterns in pre-term and term infants. Sub-scores are made up of dichotomous assessments of jaw and tongue movements during a feed. An overall sucking pattern of "normal," "disorganized," or "dysfunctional" is determined based on the items checked in each category.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie L Maitre, MD, PhD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kjeldsen CP, Neel ML, Stark AR, He Z, Chorna O, Benninger K, Maitre NL. Contingent mother's voice intervention facilitates attention in hospitalized preterm infants with neural insults. Mind Brain Educ. 2025 Feb;10(1):37-46. doi: 10.1111/mbe.70000. Epub 2025 Feb 22. PMID 40486963